CLINICAL TRIAL: NCT06193330
Title: Use of Antibiotics-cement Coated Plate in the Treatment of Gustilo-Anderson Type III Long Bone Fractures in Low- and Middle-income Countries vs External Fixation: A Multi-centre Randomized Control Trial
Brief Title: External Fixator or Antibiotic-coated Plate in Severe Open Long Bone Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oluwasegun Aremu (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor-Investigator, Oluwasegun Aremu, DR, University College Hospital, Ibadan
Organization: University College Hospital, Ibadan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: interventional
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Fracture Related Infection
MeSH Terms: interventions — External Fixators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- antibiotic-coated plate (Experimental): participants will receive antibiotic-coated plate for treatment of their type III open long bone fractures
  Interventions: Procedure: antibiotic-coated plate
- External Fixator (Active Comparator): participants will receive external fixator for treatment of their type III open long bone fractures
  Interventions: Procedure: external fixator

INTERVENTIONS:
Procedure: antibiotic-coated plate — A plate for fixing long bone fractures is coated with antibiotics cement prepared in theatre
  Arms: antibiotic-coated plate
Procedure: external fixator — external fixators are applied to participants with severe long bone fractures
  Arms: External Fixator

SUMMARY:
The purpose of the study is to assess whether infection rate is reduced with use of antibiotic-coated plate in severe open tibial fractures compare to use of external fixators

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18yrs,
* Gustilo-Anderson IIIA and IIIB open fractures,
* involvement of any long bone fractures that can be fixed with either plate or uniplanar external fixation,
* wound can be closed primarily, with skin graft or flap, or can heal secondarily

Exclusion Criteria:

* Patients with traumatic brain injury,
* spinal cord injury,
* severe burns,

  * 1 long bone fractures,
* refusal to consent,
* history of allergies to ceftriaxone or sulbactam,
* fractures associated with vascular injury
* and non-compliance with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
number of participants with fracture-related infection after 1 year | one year
  participants will be followed-up for one year and occurrence of infection at any point during this time period will be noted and recorded once

SECONDARY OUTCOMES:
number of participants who have fracture union after one year | one year
  participants will be assessed clinically and radiologically at 3months, 6months, and one year
number of participants who require re-operation after one year | one year
  during the course of follow-up, Patients with infection or other complications like malunion or non-union who require surgical intervention to achieve union will be noted and recorded
change in 12-item Short Form Survey (SF-12) score at baseline and at one year follow-up | one year
  SF-12 score of participants will be taking at baseline and also at one year of follow-up and these two scores will be assessed to determine any differences

OTHER OUTCOMES:
sub-group analysis of infection rate between smokers and non-smokers | one year
  The participants will be grouped into smokers and non-smokers and the infection rate between the two groups will be compared
sub-group analysis of infection rate between participants with and without co-morbidities | one year
  The participants will be grouped into those with co-morbidities and those without and the infection rate between the two groups will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Oluwasegun Aremu, Principal Investigator — University College Hospital, Ibadan, Nigeria
Locations (2):
- Nigeria (2):
  - Federal Medical Centre, Owo, Owo, Ondo State
  - Univeristy College Hospital, Ibadan, Nigeria, Ibadan, Oyo State

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Diwan A, Eberlin KR, Smith RM. The principles and practice of open fracture care, 2018. Chin J Traumatol. 2018 Aug;21(4):187-192. doi: 10.1016/j.cjtee.2018.01.002. Epub 2018 Feb 21. PMID 29555119
- [Background] Blease R, Kanlic E. Management of open fractures. Bosn J Basic Med Sci. 2005 Nov;5(4):14-21. doi: 10.17305/bjbms.2005.3224. PMID 16351592
- [Background] Odatuwa-Omagbemi DO. Open fractures: epidemiological pattern, initial management and challenges in a sub-urban teaching hospital in Nigeria. Pan Afr Med J. 2019 Jul 19;33:234. doi: 10.11604/pamj.2019.33.234.18141. eCollection 2019. PMID 31692766
- [Background] Ikem IC, Oginni LM, Bamgboye EA. Open fractures of the lower limb in Nigeria. Int Orthop. 2001;25(6):386-8. doi: 10.1007/s002640100277. PMID 11820448
- [Background] Conway JD, Hlad LM, Bark SE. Antibiotic cement-coated plates for management of infected fractures. Am J Orthop (Belle Mead NJ). 2015 Feb;44(2):E49-53. PMID 25658083
- [Background] Ifesanya AO, Alonge TO. Operative stabilization of open long bone fractures: A tropical tertiary hospital experience. Niger Med J. 2012 Jan;53(1):16-20. doi: 10.4103/0300-1652.99825. PMID 23271839
- [Background] Ifesanya AO, Ogundele OJ, Ifesanya JU. Orthopaedic surgical treatment delays at a tertiary hospital in sub Saharan Africa: Communication gaps and implications for clinical outcomes. Niger Med J. 2013 Nov;54(6):420-5. doi: 10.4103/0300-1652.126301. PMID 24665159
- [Background] Metsemakers WJ, Morgenstern M, McNally MA, Moriarty TF, McFadyen I, Scarborough M, Athanasou NA, Ochsner PE, Kuehl R, Raschke M, Borens O, Xie Z, Velkes S, Hungerer S, Kates SL, Zalavras C, Giannoudis PV, Richards RG, Verhofstad MHJ. Fracture-related infection: A consensus on definition from an international expert group. Injury. 2018 Mar;49(3):505-510. doi: 10.1016/j.injury.2017.08.040. Epub 2017 Aug 24. PMID 28867644
- [Derived] Aremu O, Oyewole O, Ifesanya A, Olawoye O, Ogunlade O. Use of antibiotic-cement coated plate in the treatment of Gustilo-Anderson type III long bone fractures in low- and middle-income countries vs external fixation: A multicentre randomized control trial study protocol. Injury. 2024 Aug;55(8):111637. doi: 10.1016/j.injury.2024.111637. Epub 2024 May 28. PMID 38824836